CLINICAL TRIAL: NCT01903785
Title: The Pharmacogenetic Effects of Inhaled Salbutamol on Breathing Mechanics and Cycling Performance
Brief Title: Salbutamol, Pharmacogenetics and Breathing Mechanics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: World Anti-Doping Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H09-01154-A009
Record Dates: First submitted 2013-07-08; First posted 2013-07-19 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-10

CONDITIONS: Bronchoconstriction; Inhaled Salbutamol; Cycling Performance
Keywords: exercise-induced bronchoconstriction (EIB); inhaled salbutamol; performance enhancing; cycling
MeSH Terms: interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Salbutamol (Experimental): 400ug of salbutamol (one single inhalation) will be inhaled 60min prior to the begin of a time trial. Mean power output during the following 10km time trial will be described to 1600ug salbutamol and placebo.
  Interventions: Drug: Salbutamol
- Placebo (Placebo Comparator): 400ug of placebo (one single inhalation) will be inhaled 60min prior to the begin of a time trial. Mean power output during the following 10km time trial will be described to 400ug and 1600ug salbutamol.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Salbutamol — 60 minutes prior to the start of a 10km cycling time trial on a bike ergometer, subjects will inhale either 400ug of salbutamol 1600ug of salbutamol or 400ug of placebo in a randomly assigned manner in a single dose.
  Other Names: ventolin
  Arms: Salbutamol
Drug: Placebo
  Arms: Placebo

SUMMARY:
Athletes using asthma medications called β2-agonists win a disproportionately high number of medals at Olympic Games. Due to a large variety in the genes that affect how individuals respond to β2-agonists, the investigators will look at variations in the genetic response to these medications by dividing athletes into high-responders and low-responders. The investigators will then compare athletic performance after the inhalation of β2-agonists to placebo. Furthermore, the investigators will analyze the effect of β2-agonists on breathing mechanics. Due to differences in their anatomy females may decrease the energy needed for breathing during high-intensity exercise to a greater extent compared to male athletes after the inhalation of β2-agonists.

ELIGIBILITY:
Inclusion Criteria:

* trained, experienced cyclists
* maximal oxygen consumption of at least 50ml/kg/min or 4l/min for women; and 60ml/kg/min or 5l/min for men
* athletes with and without exercise-induced bronchoconstriction

Exclusion Criteria:

* any uncontrolled heart or lung condition
* maximal oxygen consumption of less than 50ml/kg/min or 4L/min for women; and less than 60ml/kg/min or 5L/min for men
* pregnancy
* smoking

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2013-05; Primary Completion 2014-12 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The effect of inhaled salbutamol on mean power output during cycling performance in female and male athletes | Mean power output is assessed over the duration of a 10km time trial (start of time trial until completion of time trial) on a bike ergometer.
  Athletes perform a two time trials, each on a separate day. The time trials are performed 60min after the inhalation of salbutamol or placebo.
The effect of inhaled salbutamol on work of breathing (WOB) and expiratory flow limitation (EFL) in female and male athletes | WOB and EFL will be assessed during an incremental exercise test. Exercise will start at 0 Watts and will then be increased every 2.5min by 30 Watts until maximal exertion.
  EFL and WOB will be assessed with the help of an esophageal balloon and mouth pressure.

SECONDARY OUTCOMES:
The effect of inhaled salbutamol on minute ventilation in asthmatic and non-asthmatic trained, female and male cyclists | Minute ventilation will be assessed during two 10km time trials (one time trial will be started 60min after the inhalation of salbutamol, the second time trial will be started 60min after the inhalation of placebo).

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Koehle, MD, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Environmental Physiology Laboratory, University of British Columbia, Vancouver, British Columbia, Canada